CLINICAL TRIAL: NCT01899482
Title: Manual Lymphatic Drainage in Chronic Venous Insufficiency: a Randomized Controlled Trial
Acronym: MLDCVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Lisbon (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Escola Superior de Saúde Dr. Lopes Dias, Portugal (Unknown)
Responsible Party: Principal Investigator, Rute Sofia dos Santos Crisóstomo, PhD student, Technical University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SFRH/BD/62673/2009
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Venous Insufficiency
Keywords: Venous Insufficiency; Physical Therapy Techniques; Manual Lymphatic Drainage
MeSH Terms: conditions — Venous Insufficiency | interventions — Manual Lymphatic Drainage; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual Lymphatic Drainage (Experimental): One educational session in group, and 10 individual sessions of manual lymphatic drainage in lower extremity, during approximately one month.
  Interventions: Other: Manual Lymphatic Drainage; Behavioral: Education
- Control (Active Comparator): One educational session in group.
  Interventions: Behavioral: Education

INTERVENTIONS:
Other: Manual Lymphatic Drainage
  Arms: Manual Lymphatic Drainage
Behavioral: Education — Behavioral education.

SUMMARY:
The purpose of this study is to compare functional status and quality of life of a group of patients with chronic venous insufficiency treated with manual lymphatic drainage with a group not treated with manual lymphatic drainage.

Investigators hypothesized that manual lymphatic drainage can improve:

* quality of life,
* functional status,
* calf muscle strength,
* ankle range of motion,
* edema,
* severity of disease,
* and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of chronic venous insufficiency class C3-5 for Clinical-Etiological-Anatomical-Pathological classification (CEAP).

Exclusion Criteria:

* Severe cardiac insufficiency,
* Acute venous or arterial obstruction,
* Arterial insufficiency, renal insufficiency,
* Uncompensated thyroid dysfunction,
* Pregnancy, neoplastic pathology,
* Systemic or limb infection,
* Recent musculoskeletal injury in the lower limb,
* Peripheral neuropathy in the lower limb.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Assessed at baseline (no intervention), after approximately one month, with an error of three days (10 sessions of manual lymphatic drainage, for experimental group) and after approximately two months from baseline (with an error of 5 days)
  Evaluated by portuguese version of Chronic Venous Disease Quality of Life Questionnaire (CIVIQ-2).

SECONDARY OUTCOMES:
Leg edema | Assessed at baseline (no intervention), after approximately one month, with an error of three days (10 sessions of manual lymphatic drainage, for experimental group) and after approximately two months from baseline (with an error of 5 days).
  Assessed by leg perimeter.
Lower extremity symptoms | Assessed at baseline (no intervention), after approximately one month, with an error of three days (10 sessions of manual lymphatic drainage, for experimental group) and after approximately two months from baseline (with an error of 5 days).
  With Visual Analogue Scale was assessed: pain, fatigue, heaviness, itching, sKin irritation, cramps and other.
Hemodynamic evidence of severity of chronic venous disease | Assessed at baseline (no intervention), after approximately one month, with an error of three days (10 sessions of manual lymphatic drainage, for experimental group) and after approximately two months from baseline (with an error of 5 days).
  Venous reflux and anterograde flow during manual leg compression, by duplex ultrasound in femoral vein, great saphenous vein, popliteal vein and small saphenous vein.
Clinical severity of chronic venous insufficiency | Assessed at baseline (no intervention), after approximately one month, with an error of three days (10 sessions of manual lymphatic drainage, for experimental group) and after approximately two months from baseline (with an error of 5 days).
  Assessed by Venous Clinical Severity Score.
Calf muscle strength and ankle range of motion | Assessed at aseline (no intervention), after approximately one month, with an error of three days (10 sessions of manual lymphatic drainage, for experimental group) and after approximately two months from baseline (with an error of 5 days)
  Evaluated by Biodex system 3 pro isokinetic dynamometer.
Sel-reported functional status | Assessed at aseline (no intervention), after approximately one month, with an error of three days (10 sessions of manual lymphatic drainage, for experimental group) and after approximately two months from baseline (with an error of 5 days)
  Evaluated by Portuguese version of Functional Status Questionnaire (FSQ).

CONTACTS AND LOCATIONS:
Overall Officials: Paulo AS Armada-da-Silva, PhD, Principal Investigator — Faculdade de Motricidade Humana, Estrada da Costa, 1499-002 Cruz Quebrada,Portugal, Phone number: +351214149248, parmada@fmh.utl.pt
Locations (1):
- Escola Superior de Saúde Dr. Lopes Dias, Castelo Branco, Portugal

IPD SHARING:
Plan to Share IPD: Yes
http://www.archives-pmr.org/article/S0003-9993(14)01127-7/abstract